CLINICAL TRIAL: NCT03805490
Title: Italian Validation of the Forgotten Joint Score(Fjs 2015)
Brief Title: Translation, Cross Cultural Adaptation and Validation of the Italian Version of the Forgotten Joint Score in Total Knee Arthroplasty
Acronym: FJS2015
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: FJS2015
Record Dates: First submitted 2017-11-28; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Arthroplasty; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, prospective study that has the primary goal of validating the Forgotten Joint Score (FJS)

DETAILED DESCRIPTION:
This is an observational, prospective study that has the primary goal of validating the Forgotten Joint Score (FJS) as described by Behrend and Giesinger in 2012. Patients will be given two self-assessment questionnaires (WOMAC and FJS) to perform internal consistency analysis, reliability and comparability of results in a population of people undergoing total knee replacement prosthetic surgery.

Comparison of data will be done for each patient by evaluating the evolution of the postoperative period, comparing the results obtained with a well known validated score (WOMAC).

Questionnaires will be given pre-operatively, at 6 month ± 2 weeks, and 12 month ± 1 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age range between 55 and 85 years
* Italian mother-tongue
* Patients with unilateral gonarthrosis who need total knee prosthesis

Exclusion Criteria:

* Patients with orthopedic pathologies of other origin
* Patients with history of previous articular prosthetic replacement surgery on joints of the lower limb.
* Patients with history of previous major cardiovascular events
* Patients who need aids for walking
* Patients claiming that they can not submit to follow-up and therefore can not complete the study

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both gender, aged between 55 and 85 years old, Italian mother-tongue with unilateral gonarthrosis who need total knee prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-05-13 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Validating the Forgotten Joint Score. | 18 month
  Patients will be given self-assessment questionnaires Forgotten Joint Score (FJS) to perform internal consistency analysis, reliability and comparability of results in a population of people undergoing total knee replacement prosthetic surgery.
  FJS: minimum score 0 (worse outcome); maximum 100 (better outcome)

SECONDARY OUTCOMES:
BMI | 18 months
  weight and height will be combined to calculate the BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Valerio Pascale, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, MI, Italy

REFERENCES:
- [Derived] Sansone V, Fennema P, Applefield RC, Marchina S, Ronco R, Pascale W, Pascale V. Translation, cross-cultural adaptation, and validation of the Italian language Forgotten Joint Score-12 (FJS-12) as an outcome measure for total knee arthroplasty in an Italian population. BMC Musculoskelet Disord. 2020 Jan 11;21(1):23. doi: 10.1186/s12891-019-2985-2. PMID 31926561